CLINICAL TRIAL: NCT03723057
Title: Expanded Access for AG-221
Status: No longer available | Type: Expanded Access
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: AG-221
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Expanded Access; Compassionate Use
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — enasidenib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: AG-221 — Oral AG-221 administered as directed by treating physician.
  Other Names: CC-90007; Enasidenib; Idhifa

SUMMARY:
This is an expanded access program (EAP) for eligible participants designed to provide access to AG-221.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Celgene, Summit, New Jersey, United States